CLINICAL TRIAL: NCT01740921
Title: Does Glucagon-like Polypeptide 1 Improve Vascular Function and Inflammation?
Brief Title: GLP-1 and Microvascular Function in Type 2 Diabetes
Acronym: GLP-1ADDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Principal Investigator, Katarina Kos, Senior Lecturer and Honorary Consultant Physician, Royal Devon and Exeter NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 066; 10/H0106/29 (Other: Research Ethics Committee)
Record Dates: First submitted 2012-11-22; First posted 2012-12-04 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes
Keywords: GLP-1 analogues; microvascular; inflammation; fat tissue; clot structure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — Liraglutide; Diet; Caloric Restriction; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Liraglutide (Active Comparator): Liraglutide (Victoza) daily injections
  Interventions: Drug: Liraglutide
- diet (Placebo Comparator): reduction in calorie intake
  Interventions: Other: diet
- Aspirin (Placebo Comparator): Aspirin 300mg once daily
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Liraglutide — Administered once daily
  Other Names: Victoza; GLP-1 analogue
  Arms: Liraglutide
Other: diet — reduction of caloric intake to promote weight loss
  Other Names: caloric restriction
  Arms: diet
Drug: Aspirin — 300mg of Aspirin per day
  Arms: Aspirin

SUMMARY:
Some gut hormones, called incretins, stimulate insulin production in order to control sugar levels but also activate brain centres and signal to stop eating. Current administration of incretin-based therapies mimicking these gut hormones is by subcutaneous (just under the skin) injection and has been routinely available for diabetic patients for more than 4 years. It is an effective treatment for the lowering of blood glucose with an average weight loss of about 3-4kg.Recent evidence, from animal studies and limited human studies, suggests that incretins based treatments may also have beneficial effects on blood vessel function. However, it is not known whether this effect is by direct action on the blood vessel independent of an improvement of latent inflammation which is typically associated with weight loss or an anti-inflammatory effect of the incretin treatment itself. The aim of this study is to determine whether the incretin-based diabetes treatment with the GLP-1 (Glucagon-like peptide 1) analogue Liraglutide (also known as Victoza), which mimics the actions of incretins, improves blood vessel function in individuals with type 2 diabetes. It will determine whether the improvement in blood vessel function is independent of the effect of weight loss and changes in inflammation. This by the study of vascular function before and after 4 months of Victoza treatment in subjects with Type 2 diabetes in comparison with 1) participants randomized to hypo-caloric diet to achieve a similar weight loss than with Victoza and 2) participants randomized to treatment with once daily aspirin. Comprehensive assessment of blood vessel function, body fat distribution and metabolic profile at baseline and at the end of the treatment phase will be combined with assessments of inflammation markers in blood and in fat tissue biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes and an HbA1C between 7-8.5% on a stable dose of sulphonylurea and/or metformin

Exclusion Criteria:

* use of insulin
* corticosteroids
* contraceptives, tamoxifen
* methotrexate
* DPP-IV inhibitors
* pregnancy
* lactation
* endocrine disorders
* acute MI or cerebrovascular disease
* Raynaud's disease or connective tissue disease
* current or previous history of malignancy
* subjects treated with ergotamine derivatives
* unstable blood pressure for the last 3 months
* current treatment with warfarin
* subjects on any anti-inflammatory or anti-platelet agents
* history of any bleeding disorders and GI bleeds.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
change of baseline skin maximum hyperaemia at 4 months | baseline and 4 months
  laser doppler fluximetry

SECONDARY OUTCOMES:
change of baseline peripheral arterial tone at 4 months | baseline and 4 months
  ITAMAR
change of baseline endothelial-dependent vasodilation at 4 months | baseline and 4 months
  iontophoresis
change of baseline capillary density at 4 months | baseline and 4 months
  capillaroscopy

OTHER OUTCOMES:
change of baseline clot structure at 4 months | baseline and 4 months
  rigidity and elasticity of clot structure
change of baseline adipose tissue inflammation at 4 months | baseline and 4 months
  adipose tissue biopsies will be analysed for gene expression and protein content of inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Kos, MD,PhD, Principal Investigator — University of Exeter
Locations (1):
- Peninsula Clinical Research Facility, Exeter, United Kingdom

REFERENCES:
- [Background] Pastel E, McCulloch LJ, Ward R, Joshi S, Gooding KM, Shore AC, Kos K. GLP-1 analogue-induced weight loss does not improve obesity-induced AT dysfunction. Clin Sci (Lond). 2017 Mar 1;131(5):343-353. doi: 10.1042/CS20160803. Epub 2017 Jan 3. PMID 28049736